CLINICAL TRIAL: NCT06028984
Title: Self-guided Treatment for Adolescents/Adults Navigating Depression (STAND-MDD): A Randomized Controlled Trial
Brief Title: Self-guided Treatment for Depression
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Big Health Inc. (Industry)
Collaborators: Duke University (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BH-SP-01
Record Dates: First submitted 2023-08-29; First posted 2023-09-08 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Major Depressive Disorder
Keywords: Major Depressive Disorder; MDD; depression; digital therapeutic
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Intervention app (Experimental): Digitally-delivered self-guided intervention for depression accessed via mobile app
  Interventions: Device: Intervention app
- Control app (Active Comparator): An app based control condition
  Interventions: Other: Control app

INTERVENTIONS:
Device: Intervention app — An app-based intervention for depression
  Arms: Intervention app
Other: Control app — An app with non-therapeutic content
  Arms: Control app

SUMMARY:
This study will examine the efficacy and safety of a self-guided digital therapeutic app for the adjunct treatment of Major Depressive Disorder compared to a control app in adolescents and adults.

DETAILED DESCRIPTION:
This study aims to examine the efficacy of a self-guided digital therapeutic app for depression compared to a control app in individuals aged 13 and older with a diagnosis of Major Depressive Disorder. The primary outcomes are patient- and clinician-reported depression symptom severity after 5 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Positive self report screen for depression
* Participant is at least 13 years of age
* Willing and able to provide informed consent; if under 18 years of age, willing and able to provide assent, and has a legal guardian willing and able to provide consent
* Primary diagnosis of Major Depressive Disorder (MDD)
* Under the care of a United States (U.S.)-based licensed healthcare provider and willing and able to provide contact information for the provider and sign a HIPAA release that allows investigator to contact provider
* Fluent and literate in English
* Has access to a compatible device and operating system (i.e., capable of installing the app from the Google Play or Apple App Store) and regular internet access
* Located in the continental U.S., Hawaii, or Alaska, and not planning to leave the U.S. during the primary study period

Exclusion Criteria:

* Has changed or initiated psychotherapy with a mental health professional within 30 days prior to eligibility screening
* Has received certain types of psychotherapy within the last 6 months
* Has changed prescribed psychotropic medication (initiation or change in dose) within the past 30 days
* Plans to initiate or change treatment (e.g., psychotherapy, psychotropic medication, and/or other psychosocial treatment) for a mental health disorder during study intervention period
* Suicidal behavior within the past year
* Active suicide ideation with intent within the past 3 months
* Previously participated in user testing or a clinical study at Limbix Health Inc. or Big Health Inc. (such as the STAND study or Rise study), or have used a Limbix app
* Participated in any other clinical research involving an intervention or treatment within the past 60 days
* Plans to participate in any other clinical research involving an intervention or treatment during the study intervention period
* Living in the same household as another participant in the study (e.g., a sibling)
* Has a diagnosis of MDD with psychotic features or comorbid Psychotic Disorder
* Has a concurrent diagnosis of (or has been treated for) bipolar disorder I and II or severe substance use disorder within the past year
* Has treatment resistant depression
* Is employed by Big Health Inc., or is a collaborator, associate, or relation of Big Health Inc. staff
* Any condition, comorbidity, or event (other than the above) that, in the opinion of the investigator, will prevent the participant from adhering to the protocol or benefitting from the intervention, or will prevent investigators from being able to ensure safety

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 248 (Estimated)
Dates: Start 2023-10-12 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Patient Health Questionnaire (PHQ-8) | 5 weeks post-randomization
  Validated questionnaire; an 8-item scale with total scores between 0 and 24 where higher scores indicate greater severity
Montgomery-Åsberg Depression Rating Scale (MADRS) | 5 weeks post-randomization
  Validated assessment: a 10-item scale based on clinical interview with total scores between 0 and 60 where higher scores indicate greater severity

SECONDARY OUTCOMES:
Clinically important improvement based on the Patient Health Questionnaire (PHQ-8) | 5 weeks post-randomization, 1-month followup
  5 point or greater reduction in PHQ-8 score from baseline
Response based on the Patient Health Questionnaire (PHQ-8) | 5 weeks post-randomization, 1-month followup
  50% or greater reduction in PHQ-8 score from baseline
Remission based on the Patient Health Questionnaire (PHQ-8) | 5 weeks post-randomization, 1-month followup
  PHQ-8 less than 5
Global improvement assessed using the clinician-rated Clinical Global Impression Scale - Improvement (CGI-I) | 5 weeks post-randomization, 1-month followup
  A single-item measure scored between 1 and 7 where lower scores indicate greater improvement in global functioning
Clinical Global Impression - Severity (CGI-S) | 5-weeks post-randomization, 1-month followup
  A single-item measure scored between 1 and 7 where higher scores indicate greater severity of Major Depressive Disorder Symptoms
Clinically important improvement based on the Montgomery-Åsberg Depression Scale (MADRS) | 5 weeks post-randomization, 1-month followup
  10 point or greater reduction in MADRS score from baseline
Depression severity assessed with the Patient Health Questionnaire (PHQ-8) at followup | 1-, 3- and 6-month followup
  Validated questionnaire; an 8-item scale with total scores between 0 and 24 where higher scores indicate greater severity
Clinician-rated depression severity as measured by the Montgomery-Åsberg Depression Scale (MADRS) at followup | 1 month follow up
  Validated assessment: a 10-item scale based on clinical interview with total scores between 0 and 60 where higher scores indicate greater severity

CONTACTS AND LOCATIONS:
Locations (1):
- Big Health, Inc., San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No